CLINICAL TRIAL: NCT03369327
Title: Efficacy of a Fixed-Dose Combination Pill of Sofosbuvir and Daclatasvir in Treating Hepatitis C in 200 Patients Co-infected With Human Immunodeficiency Virus
Brief Title: Sofosbuvir and Daclatasvir for Treating Hepatitis C in 200 Patients Co-infected With Human Immunodeficiency Virus
Acronym: HIV200
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: RojanPharma Pharmaceutical Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95-04-159-34058
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sofosbuvir/daclatasvir (Experimental): Once daily fixed-dose combination pill of sofosbuvir and daclatasvir for 12 weeks if the patient is non cirrhotic and for 24 weeks if cirrhotic
  Interventions: Drug: sofosbuvir and daclatasvir

INTERVENTIONS:
Drug: sofosbuvir and daclatasvir — Depending on the ART received by each patient one of the fixed-dose combination pills below will be used:
  1. Daclatasvir 30 mg and sofosbuvir 400 mg
  2. Daclatasvir 60 mg and sofosbuvir 400 mg
  3. Daclatasvir 90 mg and sofosbuvir 400 mg
  Other Names: Sovodak 30/400; Sovodak 60/400; Sovodak 90/400

SUMMARY:
In a multi-center study 200 patients co-infected with hepatitis C virus (HCV) and human immunodeficiency virus (HIV) will be treated with a fixed-dose combination pill combined of 400 mg sofosbuvir and 30, 60, or 90 mg of daclatasvir - depending on the particular antiretroviral treatment (ART) being used by the patient. The treatment duration will be 12 weeks for subjects without cirrhosis and 24 weeks for those with cirrhosis.

DETAILED DESCRIPTION:
To achieve the goal of elimination of hepatitis C in 2030 as set forward by the world health organization (WHO) a main group requiring treatment are subjects co-infected with HIV. These subjects offer a particular challenge as they are receiving ART which frequently interferes with hepatitis treatment. The number of pills they are already taking also limits the compliance of these patients.

In order to evaluate the efficacy of a fixed-dose combination pill combined of 400 mg sofosbuvir and 30, 60, or 90 mg of daclatasvir - depending on the particular ART medicine being used by the patient - a multi-center study of 200 co-infected patients has been designed.

The treatment duration will be 12 weeks for subjects without cirrhosis and 24 weeks for those with cirrhosis.

The study is one of the pilots being run for hepatitis C elimination in Iran.

ELIGIBILITY:
Inclusion Criteria:

* Positive qualitative hepatitis C virus RNA test on two occasions at least 6 months apart
* Positive human immunodeficiency virus test

Exclusion Criteria:

* Heart rate < 50/min,
* Taking amiodarone
* Renal failure

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The sustained viral response rate | 12 weeks after end of treatment
  Qualitative hepatitis C virus RNA polymerase chain reaction

SECONDARY OUTCOMES:
Adverse drug events | weeks 2, 4, 8, 12 and 24
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, Study Chair — Tehran University of Medical Sciences
Locations (2):
- Iran (2):
  - Shariati Hospital, Tehran
  - Emam Hospital, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dehghan Manshadi SA, Merat S, Mohraz M, Rasoolinejad M, Sali S, Mardani M, Tabarsi P, Somi MH, Sedghi R, Tayeri K, Nikbin M, Karimi J, Sharifi AH, Kalantari S, Norouzi A, Merat D, Malekzadeh Z, Mirminachi B, Poustchi H, Malekzadeh R. Single-pill sofosbuvir and daclatasvir for treating hepatis C in patients co-infected with human immunodeficiency virus. Int J Clin Pract. 2021 Aug;75(8):e14304. doi: 10.1111/ijcp.14304. Epub 2021 May 17. PMID 33930223